CLINICAL TRIAL: NCT02877719
Title: The Effect of Poverty and Income Disparity on the Psychological WellBeing of Hong Kong Children
Brief Title: The Effect of Poverty on Psychological Well-being of Children
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW12-237
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Child
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children from low-income families: Children from low-income families were invited to fill in a set of questionnaires.
  Interventions: Other: Questionnaires
- Children from high income families: Children from high-income families were invited to fill in a set of questionnaires.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants were asked to respond to the Chinese version of the Center for Epidemiologic Studies Depression Scale for Children, the Rosenberg self-esteem scale, and the Pediatric Quality of Life Inventory.

SUMMARY:
The aim of this study is to explore the impacts of poverty and income disparity on the psychological well-being of Hong Kong Chinese children.

DETAILED DESCRIPTION:
It is well documented that poverty has a negative impact on the physiological well-being of children in the West. There is an imperative need for health care professionals to develop and evaluate interventions to promote the psychological wellbeing of children living in poverty. First, however, it is crucial to assess and understand how the impact of poverty, in particular the impact of income disparity, affects the psychological wellbeing of Hong Kong children before any intervention to promote it can be planned, developed, or evaluated. Unfortunately, while much public concern about poverty has concentrated on children's physical development, the impact of poverty and income disparity on their psychological well-being remains relatively underexplored. Because the cultural context in which they live is drastically different from that of Western children, the way that Chinese children view the nature and meaning of poverty, as well as their responses to it and to any psychosocial interventions, will in all likelihood differ considerably from those of Western children. Hence, the aim of this study is to explore the impacts of poverty and income disparity on the psychological well-being of Hong Kong Chinese children.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese pupils from Grades 5 and 6 of the elementary schools in Hong Kong
* be able to read Chinese and speak Cantonese
* had to live and go to school in the same district

Exclusion Criteria:

* Children with chronic illness or identified cognitive and learning problems

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hong Kong Chinese pupils from Grades 5 and 6 of the elementary schools in Hong Kong
Sampling Method: Probability Sample
Enrollment: 1725 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Levels of quality of life at baseline | baseline
  The quality of life of the participants will be measured by the Chinese version of the Pediatric Quality of Life Inventory (PedsQL). It has 23 items which are grouped into 4 subscales. They are physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants were asked to rate how often they had experienced problems over the past month on a scale from 0 to 4. Higher scores indicate better quality of life. Participants will be asked to respond to the Chinese version of the Pediatric Quality of Life Inventory (PedsQL) at baseline.

SECONDARY OUTCOMES:
Levels of self-esteem at baseline | baseline
  The self-esteem of the participants will be measured by the Chinese version of the Rosenberg Self-esteem Scale (RSES). It contains 10 items which are measured on a 4-point Likert scale. Each item is rated from 1 to 4. The higher scores represent the higher levels of global self-esteem of children. Participants will be asked to respond to the Chinese version of the Rosenberg Self-esteem Scale (RSES) at baseline.
Number of depressive symptoms at baseline | baseline
  The number of depressive symptoms of the participants will be measured by the Chinese version of The Center for Epidemiologic Studies Depression Scale for Children (CES-DC). It consists of 20 items that are measured on a 4-point Likert scale in relation to the experience of last week. Each item is rated from 0 to 3. The higher scores of CES-DC indicate the high numbers of depressive symptoms. The cutoff of this scale is 16, which indicates the children currently experiencing a significant level of depressive symptoms Participants will be asked to respond to the Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KY, Li WH, Chung JO, Lam KK, Chan SS, Xia W. Factors contributing to the psychological well-being for Hong Kong Chinese children from low-income families: a qualitative study. Int J Ment Health Syst. 2016 Sep 8;10(1):56. doi: 10.1186/s13033-016-0088-0. eCollection 2016. PMID 27617031